CLINICAL TRIAL: NCT00837265
Title: A Randomized Study of Subcutaneously Administered Neugranin (Recombinant Human Albumin-Human Granulocyte Colony Stimulating Factor) or Pegfilgrastim in Subjects With Breast Cancer Receiving Myelosuppressive Chemotherapy (Doxorubicin/Docetaxel)
Brief Title: Balugrastim (Neugranin) in Breast Cancer Participants Receiving Doxorubicin/Docetaxel
Acronym: NEUGR-002
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEUGR-002
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2023-02-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Breast Cancer Supportive Care Neutropenia
MeSH Terms: interventions — balugrastim; pegfilgrastim; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Pilot Phase: Balugrastim Low Dose (Experimental): Participants will receive balugrastim low dose administered by subcutaneous (SC) injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
  Interventions: Biological: Balugrastim; Drug: Chemotherapy Regimen
- Pilot Phase: Balugrastim Medium Dose (Experimental): Participants will receive balugrastim medium dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
  Interventions: Biological: Balugrastim; Drug: Chemotherapy Regimen
- Pilot Phase: Balugrastim High Dose (Experimental): Participants will receive balugrastim high dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
  Interventions: Biological: Balugrastim; Drug: Chemotherapy Regimen
- Pilot Phase: Pegfilgrastim (Active Comparator): Participants will receive pegfilgrastim 6 mg administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
  Interventions: Drug: Pegfilgrastim; Drug: Chemotherapy Regimen
- Main Phase: Balugrastim Medium Dose (Experimental): Participants will receive balugrastim medium dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
  Interventions: Biological: Balugrastim; Drug: Chemotherapy Regimen
- Main Phase: Balugrastim High Dose (Experimental): Participants will receive balugrastim high dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
  Interventions: Biological: Balugrastim; Drug: Chemotherapy Regimen
- Main Phase: Pegfilgrastim (Active Comparator): Participants will receive pegfilgrastim 6 mg administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
  Interventions: Drug: Pegfilgrastim; Drug: Chemotherapy Regimen

INTERVENTIONS:
Biological: Balugrastim — Balugrastim (Recombinant Human Albumin-Human Granulocyte Colony Stimulating Factor) will be administered per dose and schedule specified in the arm description.
  Other Names: Neugranin
  Arms: Main Phase: Balugrastim High Dose; Main Phase: Balugrastim Medium Dose; Pilot Phase: Balugrastim High Dose; Pilot Phase: Balugrastim Low Dose; Pilot Phase: Balugrastim Medium Dose
Drug: Pegfilgrastim — Pegfilgrastim will be administered per dose and schedule specified in the arm description.
  Arms: Main Phase: Pegfilgrastim; Pilot Phase: Pegfilgrastim
Drug: Chemotherapy Regimen — The chemotherapy regimen consisting of doxorubicin 60 mg/square meter (m^2) and docetaxel 75 mg/m^2 will be administered sequentially by intravenous (IV) infusion on Day 1 of treatment for up to four 21-day cycles.

SUMMARY:
Determination of the effect of balugrastim on the duration and severity of severe neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer participants scheduled to receive the AT regimen (doxorubicin/ docetaxel).

Exclusion Criteria:

* Participants may have received no more than 1 prior chemotherapy regimen (including adjuvant therapy if given within the last 12 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2008-08-21 (Actual); Primary Completion 2009-06-26 (Actual); Study Completion 2009-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Phase: Balugrastim Low Dose: Participants received balugrastim low dose administered by subcutaneous (SC) injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
- Pilot Phase: Balugrastim Medium Dose; Main Phase: Balugrastim Medium Dose: Participants received balugrastim medium dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
- Pilot Phase: Balugrastim High Dose; Main Phase: Balugrastim High Dose: Participants received balugrastim high dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
- Pilot Phase: Pegfilgrastim; Main Phase: Pegfilgrastim: Participants received pegfilgrastim 6 mg, administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
Period: Pilot Phase
Arm/Group | Pilot Phase: Balugrastim Low Dose | Pilot Phase: Balugrastim Medium Dose | Pilot Phase: Balugrastim High Dose | Pilot Phase: Pegfilgrastim | Main Phase: Balugrastim Medium Dose | Main Phase: Balugrastim High Dose | Main Phase: Pegfilgrastim
Started | 11 | 21 | 20 | 26 | 0 | 0 | 0
Modified Intent-to-treat (mITT) Population (All participants who were randomized into the study and received at least 1 dose of assigned study drug.) | 10 | 21 (1 participant was randomized to this arm but was treated with pegfilgrastim. This participant was included in the pegfilgrastim group for safety analyses.) | 20 | 25 | 0 | 0 | 0
Completed | 8 | 18 | 17 | 22 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 2 | 0 | 0 | 0
Not completed — Decision of the investigator | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant left the city | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Main Phase
Arm/Group | Pilot Phase: Balugrastim Low Dose | Pilot Phase: Balugrastim Medium Dose | Pilot Phase: Balugrastim High Dose | Pilot Phase: Pegfilgrastim | Main Phase: Balugrastim Medium Dose | Main Phase: Balugrastim High Dose | Main Phase: Pegfilgrastim
Started | 0 | 0 | 0 | 0 | 86 | 84 | 86
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 85 | 84 | 86
Completed | 0 | 0 | 0 | 0 | 76 | 79 | 83
Not Completed | 0 | 0 | 0 | 0 | 10 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2 | 1
Not completed — Decision of the investigator | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Principal investigator resignation | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Participant's personal reason | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all participants who were randomized into the study and received at least 1 dose of assigned study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Phase: Balugrastim Low Dose | Pilot Phase: Balugrastim Medium Dose | Pilot Phase: Balugrastim High Dose | Pilot Phase: Pegfilgrastim | Main Phase: Balugrastim Medium Dose | Main Phase: Balugrastim High Dose | Main Phase: Pegfilgrastim | Total
Number analyzed (Participants) | 10 | 21 | 20 | 25 | 85 | 84 | 86 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.90 (9.46) | 51.38 (10.27) | 53.75 (9.52) | 52.84 (10.36) | 49.19 (9.87) | 49.82 (9.55) | 50.26 (9.09) | 50.55 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 20 | 25 | 85 | 83 | 86 | 330
  Male | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 10 | 21 | 20 | 25 | 85 | 84 | 86 | 331

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Neutropenia in Cycle 1
Description: Severe neutropenia was defined as Grade 4 neutropenia (absolute neutrophil count [ANC] <0.5 x 10^9/liter [L]). The duration of severe neutropenia was calculated by cycle as the number of days from the first day in which the ANC fell below 0.5 x 10^9/L after beginning a chemotherapy cycle until the participant had an ANC ≥0.5 x 10^9/L within the cycle.
Time Frame: Cycle 1 (cycle length = 21 days)
Population: mITT population included all participants who were randomized into the study and received at least 1 dose of assigned study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pilot Phase: Balugrastim Low Dose | Pilot Phase: Balugrastim Medium Dose | Pilot Phase: Balugrastim High Dose | Pilot Phase: Pegfilgrastim | Main Phase: Balugrastim Medium Dose | Main Phase: Balugrastim High Dose | Main Phase: Pegfilgrastim
Number analyzed (Participants) | 10 | 21 | 20 | 25 | 84 | 84 | 86
days | 0.9 (1.37) | 1.6 (1.83) | 1.1 (1.48) | 0.9 (1.13) | 1.0 (1.09) | 1.3 (1.22) | 1.2 (1.34)

2. Secondary Outcome: Number of Participants With Febrile Neutropenia
Description: Febrile neutropenia was defined as an imputed or observed ANC <0.5 x 10^9/L and oral temperature ≥38.2 degrees celsius (°C) occurring on the same day. Number of participants with febrile neutropenia over all cycles (Cycles 1 to 4) has been reported.
Time Frame: Cycles 1 to 4 (each cycle length = 21 days)
Population: mITT population included all participants who were randomized into the study and received at least 1 dose of assigned study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Phase: Balugrastim Low Dose | Pilot Phase: Balugrastim Medium Dose | Pilot Phase: Balugrastim High Dose | Pilot Phase: Pegfilgrastim | Main Phase: Balugrastim Medium Dose | Main Phase: Balugrastim High Dose | Main Phase: Pegfilgrastim
Number analyzed (Participants) | 10 | 21 | 20 | 25 | 85 | 84 | 86
Participants | 2 | 3 | 2 | 2 | 4 | 5 | 3

3. Secondary Outcome: Duration of Severe Neutropenia in Cycles 2, 3, and 4
Description: Severe neutropenia was defined as Grade 4 neutropenia (ANC <0.5 x 10^9/L). The duration of severe neutropenia was calculated by cycle as the number of days from the first day in which the ANC fell below 0.5 x 10^9/L after beginning a chemotherapy cycle until the participant had an ANC ≥0.5 x 10^9/L within the cycle.
Time Frame: Cycles 2, 3, and 4 (each cycle length = 21 days)
Population: mITT population included all participants who were randomized into the study and received at least 1 dose of assigned study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified cycle.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pilot Phase: Balugrastim Low Dose | Pilot Phase: Balugrastim Medium Dose | Pilot Phase: Balugrastim High Dose | Pilot Phase: Pegfilgrastim | Main Phase: Balugrastim Medium Dose | Main Phase: Balugrastim High Dose | Main Phase: Pegfilgrastim
Number analyzed (Participants) | 9 | 21 | 19 | 24 | 83 | 84 | 84
days
  Cycle 2 | 0.0 (0.00) | 0.8 (1.22) | 0.4 (0.68) | 0.5 (0.88) | 0.5 (0.80) | 0.4 (0.80) | 0.5 (0.94)
  Cycle 3: number analyzed (Participants) | 8 | 20 | 18 | 24 | 82 | 81 | 84
  Cycle 3 | 0.5 (1.07) | 0.7 (0.92) | 0.6 (1.24) | 0.3 (0.61) | 0.4 (0.78) | 0.5 (1.00) | 0.4 (0.71)
  Cycle 4: number analyzed (Participants) | 8 | 18 | 17 | 22 | 79 | 79 | 84
  Cycle 4 | 0.9 (0.99) | 0.3 (0.77) | 0.1 (0.49) | 0.7 (1.25) | 0.4 (0.79) | 0.6 (1.06) | 0.6 (1.03)

4. Secondary Outcome: Time to Absolute Neutrophil Count (ANC) Recovery in Cycles 1, 2, 3, and 4
Description: Time to ANC recovery was defined as the time from the nadir ANC to an ANC ≥1.5 x 10^9/L and was calculated for participants with ANC <1.5 x 10^9/L after the beginning of a chemotherapy cycle. Time to ANC recovery was calculated by cycle as the number of days from the nadir (the lowest ANC during a chemotherapy cycle) until a participant reached an ANC >1.5 x 10^9/L.
Time Frame: Cycles 1, 2, 3, and 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pilot Phase: Balugrastim Low Dose | Pilot Phase: Balugrastim Medium Dose | Pilot Phase: Balugrastim High Dose | Pilot Phase: Pegfilgrastim | Main Phase: Balugrastim Medium Dose | Main Phase: Balugrastim High Dose | Main Phase: Pegfilgrastim
Number analyzed (Participants) | 10 | 21 | 16 | 22 | 71 | 73 | 72
days
  Cycle 1 | 3.1 (2.38) | 2.6 (1.78) | 2.0 (1.26) | 2.4 (1.59) | 2.0 (0.94) | 2.1 (1.03) | 2.6 (1.23)
  Cycle 2: number analyzed (Participants) | 3 | 14 | 12 | 17 | 54 | 57 | 55
  Cycle 2 | 1.3 (0.58) | 2.1 (1.21) | 1.9 (0.79) | 1.9 (1.20) | 1.8 (0.80) | 1.8 (1.11) | 2.1 (1.24)
  Cycle 3: number analyzed (Participants) | 7 | 13 | 9 | 15 | 52 | 51 | 56
  Cycle 3 | 2.1 (1.46) | 2.0 (1.00) | 2.2 (1.39) | 1.9 (1.06) | 1.9 (1.08) | 2.2 (1.33) | 1.8 (0.79)
  Cycle 4: number analyzed (Participants) | 7 | 13 | 7 | 13 | 43 | 52 | 53
  Cycle 4 | 2.9 (1.68) | 1.8 (0.83) | 1.3 (0.49) | 2.3 (1.49) | 1.9 (0.85) | 2.1 (1.16) | 2.1 (1.27)

ADVERSE EVENTS:
Time Frame: From the start of study drug administration through 30 days following the final dose of study drug (up to 114 days)
Description: mITT population included all participants who were randomized into the study and received at least 1 dose of assigned study drug. Per planned analysis, adverse events are reported combined for pilot and main phase.
Groups:
- Balugrastim Low Dose: Participants received balugrastim low dose administered by subcutaneous (SC) injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
- Balugrastim Medium Dose: Participants received balugrastim medium dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
- Balugrastim High Dose: Participants received balugrastim high dose administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
- Pegfilgrastim: Participants received pegfilgrastim 6 mg, administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days).
Arm/Group | Balugrastim Low Dose | Balugrastim Medium Dose | Balugrastim High Dose | Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 3/10 | 11/105 | 9/104 | 10/112
Other Adverse Events (participants affected / at risk) | 9/10 | 102/105 | 100/104 | 105/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balugrastim Low Dose (N=10) | Balugrastim Medium Dose (N=105) | Balugrastim High Dose (N=104) | Pegfilgrastim (N=112)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 7 (7) | 7 (7) | 5 (6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyclothymic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balugrastim Low Dose (N=10) | Balugrastim Medium Dose (N=105) | Balugrastim High Dose (N=104) | Pegfilgrastim (N=112)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 24 (83) | 18 (39) | 19 (56)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 4 (19) | 29 (50) | 32 (66) | 31 (71)
Lymphopenia (Blood and lymphatic system disorders) | 2 (7) | 3 (7) | 2 (2) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (12) | 59 (143) | 57 (126) | 54 (138)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 3 (8) | 3 (12) | 5 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 15 (32) | 19 (34) | 17 (31)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 4 (9) | 7 (19) | 5 (18)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (11) | 2 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 9 (9) | 14 (15) | 14 (17)
Nausea (Gastrointestinal disorders) | 4 (8) | 41 (86) | 49 (118) | 51 (121)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 8 (10) | 5 (9) | 9 (14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 11 (14) | 11 (16) | 12 (13)
Asthenia (General disorders) | 1 (2) | 30 (91) | 32 (91) | 36 (101)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 16 (38) | 16 (36) | 15 (25)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 6 (8) | 6 (6)
Respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 7 (7)
Alanine aminotransferase increased (Investigations) | 1 (2) | 4 (5) | 2 (2) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 4 (5) | 2 (2) | 3 (4)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 15 (28) | 18 (39) | 13 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (2) | 8 (14) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (18) | 17 (31) | 14 (33)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (22) | 4 (6) | 3 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (4)
Headache (Nervous system disorders) | 0 (0) | 9 (18) | 12 (27) | 14 (31)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 5 (5) | 4 (4) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (7) | 78 (79) | 68 (72) | 62 (66)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (20) | 6 (14) | 9 (20)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.